CLINICAL TRIAL: NCT03513523
Title: A Randomized, Double-Blind, Double-Dummy, Placebo-Controlled Study to Assess the Relationship Between Daily Dosing of NRPT and Changes in Liver Fat in Healthy Volunteers
Brief Title: Study to Assess the Relationship Between Daily Dosing of NRPT and Changes in Liver Fat in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elysium Health (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ELYS-170004-FL-PR
Record Dates: First submitted 2018-03-20; First posted 2018-05-01 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Fatty Liver
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: 1X dose of NRPT (Experimental): 250 mg of NR and 50 mg of PT
  Interventions: Dietary Supplement: Group 1 NRPT
- Group 2: 2X dose of NRPT (Experimental): 500 mg of NR and 100 mg of PT
  Interventions: Dietary Supplement: Group 2 NRPT
- Group 3: Placebo (Placebo Comparator): Placebo capsules contain microcrystalline cellulose, silicon dioxide and magnesium stearate
  Interventions: Other: Group 3 Placebo

INTERVENTIONS:
Dietary Supplement: Group 1 NRPT — Two capsules of NRPT and two placebo will be taken once daily in the morning for 26 weeks. Each NRPT capsule will contain 125 mg NR and 25 mg PT.
  Arms: Group 1: 1X dose of NRPT
Dietary Supplement: Group 2 NRPT — Four capsules of NRPT will be taken once daily in the morning for 26 weeks. Each NRPT capsule will contain 125 mg NR and 25 mg PT.
  Arms: Group 2: 2X dose of NRPT
Other: Group 3 Placebo — Four placebo capsules will be taken once daily in the morning for 26 weeks.
  Arms: Group 3: Placebo

SUMMARY:
The purpose of this study is to determine if there is a relationship between daily consumption of NRPT, over a six-month (26-week) period, and changes in liver fat accumulation, compared to placebo and change from Baseline in healthy volunteers. In addition, an exploratory assessment of markers of inflammation and liver fat metabolism will be examined.

ELIGIBILITY:
Inclusion Criteria:

1. MRI-PDFF of at least 15%, as measured at Visit 2 (Baseline).
2. Men or women between the ages of 18 and 70 years.
3. BMI between 25.0 and 39.9 kg/m2.
4. Non-smokers (>3 months of non-smoking).
5. If on a statin regimen, history (> 1 month) of stable dose.
6. Able to understand and cooperate with study procedures, and have signed a written informed consent prior to any study procedures.

Exclusion Criteria:

1. Diagnosis of NASH (Non-Alcoholic Steatohepatitis).
2. Bilirubin >2x ULN
3. Other causes of liver inflammation including Hepatitis A, B or C, HIV, confirmed or suspected cirrhosis, Wilson's disease, autoimmune hepatitis, hemochromatosis, alcoholic steatohepatitis, pancreatitis, or prescription medications known to cause liver damage, or known to be hepatotoxic. (Evidence of hepatocellular injury or hepatocyte ballooning.)
4. Subjects with a history of bariatric surgery.
5. Significant weight loss (> 5% body weight) or rapid weight loss (> 1.6kg/week), within six (6) months of the Screening Visit.
6. Current or recent (within six (6) months of the Screening Visit) history of significant gastrointestinal, renal, pulmonary, hepatic or biliary disease, endocrine diseases (Type II Diabetes permitted) or other invasive weight loss treatments.
7. Individual taking prescription or over-the-counter medications, including dietary supplements, known to alter lipid metabolism or liver function, within four (4) weeks of randomization.
8. Use of supplements containing pterostilbene, resveratrol, nicotinamide, or niacin, or consumption of red wine (more than 8 oz. per week) or blueberries (more than one serving per week).
9. Pregnant or lactating women or women of childbearing potential who are not using an approved method of contraception. A woman is considered to be of childbearing potential unless she is post-hysterectomy, one or more years postmenopausal, or one or more years following tubal ligation.
10. History of significant cardiovascular or coronary heart disease (CVD or CHD, respectively) as defined as having had a coronary artery bypass procedure, coronary stent or angioplasty, or myocardial infarction in the previous six (6) months.
11. History of cancer, other than non-melanoma skin cancer and basal cell carcinoma, within the previous five years.
12. Poorly controlled or uncontrolled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥95 mmHg).
13. Recent history of prolonged alcohol (>3 months) use (within past six (6) months) or excessive alcohol use, defined as >14 drinks per week (one drink = 12 oz. beer, 4 oz. wine, 1.5 oz. hard liquor).
14. Exposure to any investigational agent within four (4) weeks or five (5) half-lives, prior to the Screening Visit.
15. Subjects planning to undergo surgery during the study period or up to 1 month after the study
16. Any serious psychiatric disease or disorder, which, in the opinion of the investigator, would preclude the subject from participating in the study.
17. Any known intolerance to the investigational ingredients of this investigational product.
18. Has a condition the Investigator believes would interfere with the evaluation of the subject, or may put the subject at undue risk during the course of the study, including potentially abnormal lab results, due to a traumatic event.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Change in Fatty Liver Index | 6 months
  Change from Baseline in Fatty Liver Index (FLI) will be evaluated within each subject and compared between treatment groups.
  FLI: = (e^0.953*loge (triglycerides) + 0.139*BMI + 0.718*loge (GGT) + 0.053*waist circumference - 15.745) / (1 + e^0.953*loge (triglycerides) + 0.139*BMI + 0.718*loge (GGT) + 0.053*waist circumference - 15.745) * 100.
Change in Hepatic Fat Fraction | 6 months
  Change from Baseline in mean percent HFF across all nine Couinaud segments will be evaluated within each subject and compared between treatment groups.
Change in Insulin Resistance (HOMA-IR) | 6 months
  Change from Baseline in HOMA-IR will be evaluated within each subject and compared between treatment groups.
  HOMA-IR: = ([glucose x insulin]/450) For this measure, the comparison is between the placebo and the two IP groups at end-of-study
Change in liver fat content | 6 months
  To determine if there is a dose effect of NRPT on changes from baseline in liver fat content compared to placebo, as determined by MRI-PDFF.

SECONDARY OUTCOMES:
Safety: Adverse Events | 6 months
  To determine the safety of NRPT as measured by number of adverse events and serious adverse events.
Safety: LFT's | 6 months
  To determine the safety of NRPT as measured by change in liver function tests (AST U/L, ALT U/L, GGT U/L, Alk Phos U/L) from baseline.

OTHER OUTCOMES:
Exploratory: Change in Inflammatory Marker (hsCRP) | 6 months
  Change from Baseline in hsCRP will be evaluated within each subject and compared between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Chen, PhD, Principal Investigator — Biofortis Clinical Research, Inc.
Locations (9):
- United States (9):
  - Indago Research and Health Center, Hialeah, Florida
  - Altus Research, Inc., Lake Worth, Florida
  - Lone Star Research Center, Miami, Florida
  - Med-Care Research Corp, Miami, Florida
  - Legacy Clinical Solutions: Sensible Healthcare, LLC, Ocoee, Florida
  - IMIC, Inc, Palmetto Bay, Florida
  - Lenus Research & Medical Group, Sweetwater, Florida
  - Barrett Clinic, P.C., La Vista, Nebraska
  - Trial Management Associates, LLC, Wilmington, North Carolina

REFERENCES:
- [Derived] Dellinger RW, Holmes HE, Hu-Seliger T, Butt RW, Harrison SA, Mozaffarian D, Chen O, Guarente L. Nicotinamide riboside and pterostilbene reduces markers of hepatic inflammation in NAFLD: A double-blind, placebo-controlled clinical trial. Hepatology. 2023 Sep 1;78(3):863-877. doi: 10.1002/hep.32778. Epub 2022 Nov 22. PMID 36082508